CLINICAL TRIAL: NCT01813175
Title: Randomised, Controlled, Double-blind Exploratory Study to Investigate the Effect of Specific Synbiotics Mixtures on Gut Microbiota Composition in Healthy Infants.
Brief Title: Color Synbiotics Study
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Danone Asia Pacific Holdings Pte, Ltd. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Other
Other Study IDs: COL.1.C.A
Record Dates: First submitted 2013-03-12; First posted 2013-03-18 (Estimated); Last update posted 2017-09-07 (Actual); Status verified 2017-09

CONDITIONS: Beneficial Bacteria in Gut

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator
Oversight: Data Monitoring Committee: No

ARMS (4):
- Intervention Group I (Active Comparator): Regular non-hydrolysed cow's milk based infant formula with synbiotics mixture I
  Interventions: Other: Regular non-hydrolysed cow's milk I
- Interventional Group II (Active Comparator): Regular non-hydrolysed cow's milk based infant formula with synbiotics mixture II
  Interventions: Other: Regular non-hydrolysed cow's milk II
- Control Group (Placebo Comparator): Regular non-hydrolysed cow's milk based infant formula
  Interventions: Other: Regular non-hydrolysed cow's milk - control
- Reference Group (No Intervention): Exclusively breast-fed infants

INTERVENTIONS:
Other: Regular non-hydrolysed cow's milk I — Regular non-hydrolysed cow's milk based infant formula with synbiotics mixture I
  Arms: Intervention Group I
Other: Regular non-hydrolysed cow's milk II — Regular non-hydrolysed cow's milk based infant formula with synbiotics mixture II
  Arms: Interventional Group II
Other: Regular non-hydrolysed cow's milk - control — Regular non-hydrolysed cow's milk based infant formula without synbiotics mixture
  Arms: Control Group

SUMMARY:
This study is initiated to investigate the effect of infant formula with added specific synbiotics mixture on proportion of beneficial bacteria.

ELIGIBILITY:
Inclusion Criteria:

* Healthy term infants (gestational age ≥ 37 1/7 and ≤ 41 6/7 weeks) aged 46 - 65 days (inclusive) at entry into the study
* Fully formula fed for at least one week (not applicable for the breastfeeding reference group since these infants must be exclusively breastfed before and throughout the study)
* Parents' or legal guardian's written informed consent

Exclusion Criteria:

* Exclusion criteria for run-in period (visit 1, screening) are:
* Being weaned before inclusion (introduction of any other foods other than formula or human milk)
* Moderate or severe acute malnutrition, defined as weight-for-age and sex below -2 z-scores of the median WHO growth standards
* Medical condition for which a special diet other than standard (non hydrolised) cow's milk-based infant formula is required
* Known congenital diseases or malformations which could interfere with the study (e.g. gastrointestinal malformations, congenital immunodeficiency), as per investigator's clinical judgement
* Use of systemic antibiotics or anti-mycotic drugs in the 4 weeks prior to entry into the study
* Received Inactivated Poliovirus Vaccine (IPV) or Rotavirus Vaccine (RV) prior to entry into the study
* Gastroenteritis or diarrhoea in the last two weeks prior to entry into the study
* Participation in any other studies involving investigational or marketed products concomitantly or within two weeks prior to entry into the study
* Investigator's uncertainty about the willingness or ability of the parents to comply with the protocol requirements

Ages: 43 Days to 65 Days | Sex: All | Healthy Volunteers: Yes
Age Groups: Child
Enrollment: 290 (Actual)
Dates: Start 2013-05; Primary Completion 2016-07 (Actual); Study Completion 2016-07 (Actual)

PRIMARY OUTCOMES:
Change of Baseline proportion of beneficial bacteria at week 6 in interventional group compared to the change in control group | baseline, week 6

SECONDARY OUTCOMES:
Change of proportion of baseline beneficial bacteria at week 6 in interventional group I compared to the change in control group | baseline, week 6
Change of Baseline proportion of beneficial bacteria at week 6 in interventional group II compared to the change in control group | baseline, week 6

CONTACTS AND LOCATIONS:
Locations (3):
- Thailand (3):
  - Thammasat Hospital, Klong Luang, Changwat Pathum Thani
  - King Chulalongkorn Memorial Hospital, Bangkok
  - Phramongkutklao Hospital, Bangkok

REFERENCES:
- [Derived] Phavichitr N, Wang S, Chomto S, Tantibhaedhyangkul R, Kakourou A, Intarakhao S, Jongpiputvanich S; COLOR Study Group; Roeselers G, Knol J. Impact of synbiotics on gut microbiota during early life: a randomized, double-blind study. Sci Rep. 2021 Feb 11;11(1):3534. doi: 10.1038/s41598-021-83009-2. PMID 33574421